CLINICAL TRIAL: NCT03274024
Title: The Asia Primary Tube Versus Trab (TVT) Study
Acronym: TVT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore Eye Research Institute (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Dr Ho Ching Lin, Research Director, Singapore Eye Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R1293/99/2015
Record Dates: First submitted 2017-08-29; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy; Mitomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tube implant (Experimental): Ahmed Glaucoma Implant (AGI) surgery
  Interventions: Device: Ahmed Glaucoma Implant
- Trabeculectomy (Active Comparator): Trabeculectomy with mitomycin C surgery
  Interventions: Procedure: Trabeculectomy with Mitomycin C

INTERVENTIONS:
Device: Ahmed Glaucoma Implant — Conjunctival Flap Scleral Exposure Insertion of Episcleral Plate Priming of the tube prior to AC entrance Insertion of Tube into the Anterior Chamber Suturing tube Coverage of tube
  Arms: Tube implant
Procedure: Trabeculectomy with Mitomycin C — Conjunctival Flap Mitomycin C Application Scleral Flap Paracentesis Excision of Limbal Tissue Peripheral Iridectomy Scleral Flap Closure Conjunctival Flap Closure
  Arms: Trabeculectomy

SUMMARY:
Comparison of Ahmed Glaucoma Implant (AGI) against trabeculectomy with mitomycin C in patients with uncontrolled open angle glaucoma

DETAILED DESCRIPTION:
The objective of the Asia Primary Tube versus Trab (TVT) study is to compare the efficacy and safety of placement of an Ahmed Glaucoma Implant (AGI) (New World Medical Inc., Rancho Cucamonga, CA, USA) against trabeculectomy with mitomycin C in patients with uncontrolled glaucoma, who may or may not have had previous clear corneal cataract surgery with intraocular lens implantation, over 5 years. Outcome discrimination between the two treatment groups will be made using following parameters:

1. Intraocular pressure
2. Need for supplemental medical therapy
3. Incidence of short and long term surgical complications and need for re-operation.
4. Visual function (Visual acuity and Visual field)

Hypothesis: Glaucoma drainage implants have better surgical outcomes in terms of IOP lowering efficacy compared to trabeculectomy with mitomycin-C over 5 years in Asian patients with medically uncontrolled glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Open angle glaucoma including primary open angle glaucoma, pseudoexfoliative or pigmentary glaucoma.
2. IOP > 18 mm Hg on 2 or more medications on at least 2 visits
3. Informed consent given and consent form signed.

Exclusion Criteria:

1. Unwilling or unable to give consent, unwilling to accept randomisation, or unable to return for scheduled protocol visits.
2. Pregnant or nursing women
3. No light perception vision
4. Previous incisional intraocular surgery, other than uncomplicated clear corneal cataract surgery
5. Previous ocular laser in study eye (keratorefractive surgery and cyclodestructive procedure), except for laser trabeculoplasty procedures (Argon Laser and Selective Laser Trabeculoplasty)
6. Iris neovascularisation or proliferative retinopathy
7. Primary angle closure or primary angle closure glaucoma
8. Iridocorneal endothelial syndrome or anterior segment dysgenesis
9. Epithelial or fibrous downgrowth
10. Aphakia
11. Chronic or recurrent uveitis
12. Severe posterior blepharitis
13. Unwilling to discontinue contact lens use after surgery
14. Glaucoma secondary to penetrating keratoplasty, trauma, steroids, retinal disease/surgery or neovascular disease
15. Conjunctival scarring from prior ocular surgery, trauma or cicatrizing disease precluding a superior trabeculectomy
16. Need for glaucoma surgery combined with other ocular procedures (i.e. cataract surgery, penetrating keratoplasty, or retinal surgery) or anticipated need for urgent additional ocular surgery
17. Advanced glaucoma with MD <-20dB

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-09-28 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Failure | 6 months
  Failure defined by ANY of the following criteria:
  * IOP ≥ 18 mm Hg on two consecutive follow-up visits after 6 months
  * IOP not reduced to 20% below baseline on two consecutive visits after 6 months
  * IOP ≤ 5 mm Hg with visually significant hypotony maculopathy on two consecutive visits after 3 months
  * Additional glaucoma surgery, excluding laser suture lysis, removal of releasable trabeculectomy or conjunctival sutures, needling of the bleb or tube plate with or without 5FU, subconjunctival 5FU injections and anterior chamber reformation.
  * Loss of light perception vision

SECONDARY OUTCOMES:
IOP | 60 months
  Intraocular pressure (mmHg)
Best Corrected Visual Acuity (BCVA) | 60 months
  ETDRS visual acuity chart (logMAR or equivalent)
Supplemental medication | 60 months
  Number of supplemental glaucoma medications used at Month 60
Adverse Events | 60 months
  Number of Adverse Events during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Ching Lin Ho, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore